CLINICAL TRIAL: NCT01287858
Title: A Phase 1, Randomized, Double Blind, Placebo Controlled, Sequential, Ascending Single-Dose and Multiple-Dose First-in-Human Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AC430 in Healthy Subjects
Brief Title: Study to Assess Safety, Tolerability, and Pharmacokinetics of Oral Doses for AC430 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC430-001
Record Dates: First submitted 2011-01-12; First posted 2011-02-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: AC430
- AC430 (Active Comparator): AC430
  Interventions: Drug: AC430

INTERVENTIONS:
Drug: AC430 — Healthy volunteers will either receive AC430 or placebo.

SUMMARY:
AC430 will be administered, orally under fasting conditions (fasting 4 hours before and 2 hours after dosing) with approximately 240 mL of water either once daily or twice daily. It is designed to assess the safety, tolerability, and pharmacokinetics of single and multiple oral doses of AC430.

DETAILED DESCRIPTION:
A dose-finding study of AC430 in healthy volunteers.

ELIGIBILITY:
Important Inclusion Criteria:

1. Healthy normal males and females, age 18 to 45, inclusive, at the time of consent
2. Able to communicate effectively in the English language
3. Able to provide valid, written informed consent
4. Able to swallow up to 20 capsules of study drug
5. BMI (body mass index) ranging between 18 and 30 kg/m2, inclusive
6. Minimum weight of 50 kg
7. Serum Creatinine ≤ ULN (upper limit of normal) and estimated creatinine clearance at screening of ≥ 80 mL/min per the Cockcroft-Gault equation
8. Total serum bilirubin ≤ ULN (may be repeated to confirm eligibility)
9. Serum aspartate transaminase (AST) and alanine transaminase (ALT) ≤ ULN (may be repeated to confirm eligibility)
10. Male subjects must either be sterile or agree to use from Check-in until 90 days following the last dose of AC430, an acceptable form of birth control.
11. Female participants must be either of non-child-bearing potential or agree to use an acceptable form of birth control.

Important Exclusion Criteria:

1. History of clinically significant drug allergy
2. Participation in another clinical trial with receipt of an Investigational Product within 90 days before dose administration (or 5 half-lives, whichever is longer)
3. Major surgery within 90 days before study enrollment
4. Use of prescription, over the counter, or herbal medications or supplements, including oral contraceptives within 14 days of check-in
5. A history of drug abuse or a history of alcohol abuse within 1 year prior to Screening
6. Current or recent (within 30 days before enrollment) use of tobacco or nicotine products
7. Consumption of alcohol containing beverages > an average of 14 drinks per week or unwillingness to refrain from ethanol consumption while confined to the study unit
8. Inadequate venous access that would interfere with obtaining blood samples
9. Recipients of blood transfusion or transfusion of blood or plasma products, within 90 days before study drug administration
10. Donation of blood ≥ 500 mL within 2 months before study drug administration
11. History or positive laboratory evidence of Human immunodeficiency virus (HIV), Hepatitis B antigen and antibody, or Hepatitis C, or history of Tuberculosis (TB) infection, or a positive result for Quantiferon Gold test
12. Prolonged average of the corrected QTc by Fridericia's correction factor (QTcF) interval on screening electrocardiogram (ECG) triplicate (≥ 450 ms for males and ≥ 470 ms for females)
13. Abnormal laboratory values that are considered clinically significant by the Investigator
14. History of cancer
15. History of eating disorders within the past 3 months
16. History of a seizure disorder or clinically significant head injury
17. Positive urine drug screen for drugs of abuse including alcohol
18. Active infection within 90 days of check-in
19. Medical condition, serious intercurrent illness, cardiovascular, pulmonary, neurologic, psychiatric, renal, hepatic or gastrointestinal disease, or other extenuating circumstance that, in the judgment of the Principal Investigator, could jeopardize subject safety or interfere with the objectives of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Assess the safety, tolerability, and pharmacokinetics of single and multiple oral doses of AC430. | 6 months
  * Number of participants with adverse events as measurement of safety and tolerability of AC430. [Time frame: 1-28 days]
  * Maximum concentration (Cmax) for AC430 in plasma (measured in ng/mL) [Time frame: 1-28 days]
  * Tmax = Time of maximum concentration of AC430 in plasma (hr) [Time frame: 1-28 days]
  * AUC = Area under the curve from the time of dosing extrapolated to infinity (ng.hr/mL) [Time frame: 1-28 days]
  * Urine: amount of AC430 excreted in urine (Ae0-48), renal clearance (CLr) and fraction of drug excreted in urine (Fe). [Time frame: 1-28 days]

SECONDARY OUTCOMES:
Determine the pharmacodynamic effects of single and multiple oral doses of AC430. | Measured at specific timepoints prior to and following dosing regimen.
  * Single ascending dose (SAD): Pharmacodynamics (blood analysis) of AC430 [Time Frame: up to 8 days post dose] [Designated as safety issue: No]
  * Multiple ascending doses (MAD): Pharmacodynamics (blood analysis) of AC430 [Time Frame: up to 17 days postdose] [Designated as safety issue: No]

CONTACTS AND LOCATIONS:
Overall Officials: Guy Gammon, MB BS, MRCP, Study Director — Interim Chief Medical Officer / Ambit Biosciences Corporation
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States